CLINICAL TRIAL: NCT05789524
Title: A Global, Open-label, Adaptive Design Study to Investigate the Efficacy and Safety of SerpinPC in Subjects with Severe Hemophilia a or Moderately Severe to Severe Hemophilia B
Brief Title: The Efficacy and Safety of SerpinPC in Participants with Severe Hemophilia a or Moderately Severe to Severe Hemophilia B
Acronym: PRESent-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to business and strategic decision
Sponsor: ApcinteX Ltd (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP-0102; 2022-502880-39-00 (Other: EU CT Number)
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hemophilia a; Hemophilia B
Keywords: SerpinPC; Hemophilia
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Protein C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 - Cohort 1: SerpinPC (Experimental): Participants will receive SerpinPC 1.2 mg/kg SC Injection QW for 24 weeks after a minimum of 12 weeks of a prospective observation period.
  Interventions: Drug: SerpinPC
- Part 1 - Cohort 2: SerpinPC (Experimental): Participants will receive SerpinPC 1.2 mg/kg SC Injection Q2W for 24 weeks after a minimum of 12 weeks of a prospective observation period.
  Interventions: Drug: SerpinPC
- Part 1 - Cohort 3: SerpinPC (Experimental): Participants will receive SerpinPC 1.2 mg/kg SC Injection Q4W for 24 weeks after a minimum of 12 weeks of a prospective observation period.
  Interventions: Drug: SerpinPC
- Part 2 - SerpinPC (Dose-confirmatory phase) (Experimental): After a minimum of 24 weeks of prospective observation, participants will receive SerpinPC at dose of 1.2 mg/kg Q2W for 24 weeks in Part 2, unless the Interim Analysis (IA) shows a greater benefit-risk profile with either the 1.2 mg/kg QW or Q4W treatment regimens.
  Interventions: Drug: SerpinPC
- Part 3 - SerpinPC (Extension phase) (Experimental): After completion of dosing in Part 1 or Part 2, participants will continue treatment with SerpinPC at the dose of SerpinPC selected for Part 2 in a 24-week extension phase (Part 3).
  Interventions: Drug: SerpinPC

INTERVENTIONS:
Drug: SerpinPC — Administered as SC injection.
  Other Names: Activated Protein C (APC) inhibitor

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, tolerability and pharmacokinetics of prophylactic SerpinPC administered subcutaneously (SC) to participants with severe hemophilia A (HemA) (with or without inhibitors) or moderately severe to severe hemophilia B (HemB) (without inhibitors) as part of the SerpinPC registrational program.

This study consists of 3 parts: Part 1: dose-justification phase, Part 2: dose-confirmatory phase, Part 3: extension phase for participants who complete either Part 1 or Part 2.

This adaptive design study has a randomized dose-justification component to investigate the efficacy and safety of SerpinPC as a therapeutic option, principally for participants with HemB without inhibitors. SerpinPC has a novel mechanism of action compared with marketed treatments and those that are in development.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants ≥12 and ≤65 years of age at the time of informed consent. Enrollment of adolescents (aged ≥12 to <18 years) will be deferred until at least 12 adult participants from each SerpinPC treatment regimen have completed at least 12 weeks of dosing in Part 1 and safety of SerpinPC has been assessed
2. Capable of providing written informed consent (adolescent assent and parental/guardian/legal representative consent when appropriate) for participation and having the opportunity to discuss the study with the investigator or delegate
3. Historically documented severe HemA (defined as factor VIII less than (<) 0.01 international unit (IU)/milliliter(mL) [<1%]), with or without inhibitors, or moderately severe to severe HemB (defined as factor IX ≤0.02 IU/mL [≤2%]), without inhibitors high titer inhibitor (high titer inhibitor defined as ≥5
4. Participant is currently included in a prophylaxis program. Fulfillment of this criterion will be based on investigator's judgment of adequate prophylaxis regimen OR participant is undergoing an on-demand treatment regimen and must have had greater than or equal to (≥) 6 documented acute bleeding episodes (spontaneous or traumatic) that required treatment during the 6 months before screening. Irrespective of the treatment program that the participant is currently undergoing, they must be willing to remain in the same program for the duration of the prospective observational period
5. Participants who are currently in a prophylaxis program must be willing to stop prophylaxis (including episodic prophylaxis for sporting events) before the first dose of SerpinPC
6. For Part 1: At least 12 weeks of prospective documentation of bleeding episodes in the AP-0105 non-interventional study before SerpinPC dosing, or willing to complete a 12-week observational period (at minimum) in AP-0102
7. For Part 2: At least 24 weeks of prospective documentation of bleeding episodes in the AP-0105 non-interventional study before SerpinPC dosing or willing to complete a 24-week observational period (at minimum) in AP-0102
8. No bleeding in the 7 days before baseline (the prospective observation period can be extended by 10 days if there is an ongoing active bleed)
9. D-dimer of less than or equal to (≤) 750 micrograms(μg)/Liter(L). In cases where there is a resolving bleed, the exclusion threshold is ≤1750 milligrams(mg)/L at Screening and Pre-dosing visits
10. Adequate hematologic function, defined as a platelet count of ≥100,000/microliters(μL) (≥100 × 109/L) and hemoglobin level of ≥10 grams(g)/deciliter(dL) (≥100 g/L or ≥6.206 millimols(mmol)/L) at Screening and Pre-dosing visits
11. Adequate hepatic function, defined as a total bilirubin level of ≤1.5*upper limit of normal (ULN) (excluding Gilbert syndrome) and aspartate aminotransferase and/or alanine aminotransferase of ≤3 × ULN at Screening and Pre-dosing visits; no clinical signs or known laboratory or radiographic evidence consistent with cirrhosis of the liver
12. Adequate renal function, defined as a serum creatinine level of ≤2.0*ULN at Screening and Pre-dosing visits
13. Able to use a diary to document bleeding events and medication usage
14. Sexually active participants with a partner who could become pregnant should agree to use effective contraception for the duration of the study effective contraceptive measures include condom with or without spermicide, a combination of male condom with either cap, diaphragm, or sponge with spermicide (double barrier methods), vasectomy, partner using stable contraceptive measures (combined [estrogen and progestogen-containing] hormonal contraception or progestogen-only hormonal contraception initiated 2 or more menstrual cycles prior to screening, intrauterine device [IUD], intrauterine hormone-releasing system [IUS], bilateral tubal ligation), and/or sexual abstinence.

Exclusion Criteria:

1. Known severe thrombophilia (defined as antithrombin deficiency and/or protein S deficiency and or protein C deficiency).
2. Participant with previous factor VIII or factor IX inhibitor who responded to immune tolerance induction and remains on prophylactic factor concentrate
3. Previous deep vein thrombosis, pulmonary embolism, myocardial infarction, or stroke
4. History of intolerance to SC injections
5. Uncontrolled hypertension (systolic blood pressure >160 millimeter of mercury (mm Hg); diastolic blood pressure >100 mm Hg)
6. Weight >150 kg OR body mass index >40 Kilograms(kg)/meter square (m2)
7. Has active cancer and/or requires therapy for cancer, except for basal cell carcinoma
8. Participation in another clinical trial (except for AP-0105) during the 30 days before Screening
9. Use of emicizumab in the 24 weeks before Baseline (Day 0)
10. Prior, ongoing, or planned treatment with gene therapy for hemophilia
11. Any major medical, psychological, or psychiatric condition that could cause the participant to be unsuitable for the study or could interfere with the interpretation of the study results
12. History of or other evidence of recent alcohol or drug abuse as determined by the investigator (in the 12 months before Screening)
13. Known human immunodeficiency virus (HIV) infection with CD4 count (or T-cell count) of <200 cells/μL within 24 weeks before Screening and Pre-dosing visits. Participants with HIV infection who have CD4 >200 and meet all other criteria are eligible
14. Current or planned treatment with anticoagulant or antiplatelet drugs
15. Is planning to donate/bank sperm during SerpinPC treatment AND within 30 days of last dose of SerpinPC
16. Any other significant conditions or comorbidities that, in the opinion of the investigator, would make the participant unsuitable for enrollment or could interfere with participation in or completion of the study

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) for Treated Bleeds up to Week 24 | Up to Week 24

SECONDARY OUTCOMES:
Annualized Bleeding Rate (ABR) for Treated Bleeds Up to Week 48 | Up to Week 48
Annualized Bleeding Rate (ABR) for Treated Spontaneous Bleeds | Up to Week 48
Annualized Bleeding Rate (ABR) for Treated Spontaneous Joint Bleeds | Up to Week 48
Total Coagulation Factor and/or Bypass Product Consumption During Parts 2 and 3 | Up to Week 48
Pharmacokinetic Plasma Concentrations of SerpinPC | From Day 1 up to 24 weeks
Haemophilia-specific QoL Instrument for Adults (Haem-A-QoL) Physical Health scale in participants aged 17 to ≤65 years with hemophilia | From Baseline up to 24 weeks
  The Haem-A-QoL instrument contains 44 items across 10 domains relevant to HRQoL in adults (physical health, feelings, view of participant's self, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership, and sexuality). Each item is rated on a 5-point scale (1=never, 2=rarely, 3=sometimes, 4=often, 5=all the time). Higher scores are indicative of greater impairment in HRQoL.
Number of Participants With Adverse Events (AEs) | From Baseline up to Week 48

CONTACTS AND LOCATIONS:
Locations (59):
- United States (10):
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Indiana Hemophilia and Thrombosis Center, Inc., Indianapolis, Indiana
  - University of Iowa Healthcare, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - East Carolina Univeristy, Greenville, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at Houston-Gulf States HTC, Houston, Texas
- Yeolyan Hematology and Oncology Center, MoH of Armenia CJSC, Yerevan, Yerevan, Armenia
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (2):
  - Queen Fabiola Children, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
- Canada (3):
  - Hamilton Health Sciences Corporation, Hamilton, Hamilton
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Unity Health Toronto, Toronto
- France (3):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, France
  - Hopital Necker - Enfants Malades, Paris, IDF
  - Hospices Civils de Lyon (HCL) - Hopital Femme-Mere-Enfant (HFME), Lyon, Rhone
- Germany (3):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Klinik fur Angiologie Hamostaseologie Haus 12 A Gerinnungssprechstunde, Berlin, State of Berlin
- India (2):
  - K J Somaiya Super Speciality Hospital & Research Centre, Mumbai, Maharashtra
  - Christian Medical College & Hospital, Ludhiana, Punjab
- Italy (5):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, MI
  - A.O.U Citt della Salute e della Scienza di Torino, Torino, Torino
  - Presidio Ospedaliero Universitario S. Maria della Misericordia - ASUFC, Udine, UD
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona, Verona
  - Azienda Ospedaliero-Universitaria Careggi, Florence
- Poland (2):
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów, Podkarpackie Voivodeship
  - Kl Hemat Now Krwi i Trans USK, Wroclaw, Woj. Dolnośląskie
- Phoenix Pharma Pty Ltd, Port Elizabeth, Eastern Cape, South Africa
- Spain (5):
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitari Vall d'Hebron, Barcelona, Spain
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga Hospital Carlos Haya - Hospital Materno-Infantil, Málaga
- Taiwan (4):
  - Taipei Veterans General Hospital, Taipei, Taipei
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (6):
  - Ege University Medical Faculty Pediatric Hospital, Izmir, İzmir
  - Trakya University Haematology Clinic, Edirne
  - Istanbul University Oncology Institute, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Izmir
  - Ege University Hospital Internal Disease, Izmir
  - Ondokuz Mayis University Medical Faculty, Samsun
- United Kingdom (10):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, Birmingham
  - University Hospital of Wales, Cardiff, Cardiff
  - Glasgow Royal Infirmary, Glasgow, Glasgow
  - Kent Canterbury Hospital, Canterbury, Kent
  - Barts and London School of Medicine and Dentistry, London, London
  - Royal Free London NHS Foundation Trust, London, London
  - Imperial College Healthcare NHS Trust, London, London
  - Oxford University Hospital, Oxford, Oxfordshire
  - Southampton General Hospital, Southampton, Southampton
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No